CLINICAL TRIAL: NCT04297098
Title: Pain Sensitivity Evaluation in Respiratory Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Marie Carmen Valenza, Universidad de Granada
Other Study IDs: DF0090UG
Record Dates: First submitted 2020-02-21; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Asthma; Pain, Chronic; Allergy
MeSH Terms: conditions — Asthma; Chronic Pain; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthmatic patients
- Allergic patients
- Control group

SUMMARY:
Previous studies have reported that asthmatic or chronic pulmonary obstructive disease patients have an increased response to pain stimulus. However, this aspect has not been evaluated in allergic patients. Additionally, the difference in pain sensitivity between asymptomatic period crisis have not been evaluated yet.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age.
* Accepted to sign the informed consent.
* Diagnosis of asthma or allergy.

Exclusion Criteria:

* Cognitive impairment.
* Orthopedic pathologies limiting test performance.
* Active smokers.
* Neurologic pathologies limiting voluntary mobility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were between 18 and 65 years of age, accepted to sign the informed consent and presented a diagnosis of persistent asthma, in a well-controlled phase, were recruited from the Pneumology Service of the "Complejo Hospitalario Universitario" (Granada).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-24 (Estimated); Primary Completion 2020-05-12 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threslhold | Baseline
  The pain pressure thresholds (PPTs) were evaluated by an analogic manual mechanical algometer. This tool consisted of a circular platform with an area of 1 cm2 area, which was perpendicularly applied to generate progressive pressure on the skin at a 1 kg/sec rate. The points selected were chose based on a previous study in asthma patients. Patient was assessed in a seated position and pressure was applied two times at five bilateral points of the body: At two distal points, the distal thumb phalangeal and the gracilis muscle tendon at the inside of the knee. Further at three points at the chest, the costae II, distal of the midst part of the clavicle, the supraspinous muscle and the trapezius muscle's second portion, between the angulus superior at scapulae and the vertebral column.
Pressure pain threslhold | Up to 24 weeks
  The pain pressure thresholds (PPTs) were evaluated by an analogic manual mechanical algometer. This tool consisted of a circular platform with an area of 1 cm2 area, which was perpendicularly applied to generate progressive pressure on the skin at a 1 kg/sec rate. The points selected were chose based on a previous study in asthma patients. Patient was assessed in a seated position and pressure was applied two times at five bilateral points of the body: At two distal points, the distal thumb phalangeal and the gracilis muscle tendon at the inside of the knee. Further at three points at the chest, the costae II, distal of the midst part of the clavicle, the supraspinous muscle and the trapezius muscle's second portion, between the angulus superior at scapulae and the vertebral column.

SECONDARY OUTCOMES:
Leicester Cough Questionnaire | Baseline
  The Leicester Cough Questionnaire (LCQ) was used to evaluate cough. This questionnaire brief, easy to administer and well-validated. It consists of 19 items with scores ranging from 1 to 7 and it is divided in three subscales: physical, psychological, and social. The minimum and maximum achievable LCQ total scores are 3 and 21, respectively. A lower LCQ score signifies more cough
Leicester Cough Questionnaire | Up to 24 weeks
  The Leicester Cough Questionnaire (LCQ) was used to evaluate cough. This questionnaire brief, easy to administer and well-validated. It consists of 19 items with scores ranging from 1 to 7 and it is divided in three subscales: physical, psychological, and social. The minimum and maximum achievable LCQ total scores are 3 and 21, respectively. A lower LCQ score signifies more cough
Borg scale | Baseline
  The Borg scale was used to assess the dyspnea, which is a comprehensive instrument designed to measure breathlessness in patients with respiratory pathology. Patients rated their dyspnoea from 0 to 10, where 0 represents "no dyspnoea" and 10 represents "maximum dyspnoea." A difference of 0.9 units was considered as the minimal clinically important difference (MCID), according to previous studies in patients with respiratory disease
Borg scale | Up to 24 weeks
  The Borg scale was used to assess the dyspnea, which is a comprehensive instrument designed to measure breathlessness in patients with respiratory pathology. Patients rated their dyspnoea from 0 to 10, where 0 represents "no dyspnoea" and 10 represents "maximum dyspnoea." A difference of 0.9 units was considered as the minimal clinically important difference (MCID), according to previous studies in patients with respiratory disease
Catastrophizing about Asthma Scale | Baseline
  In the Catastrophizing about Asthma Scale (CAS) patients rate the extent to which 24 items expressing catastrophic thoughts and feelings about asthma are applicable to themselves (e.g., "There is nothing I can do to reduce the intensity of the asthma attack", "I worry all the time about whether the asthma attack will end", "I feel I can't go on"). The scale has two subscales, one referring to the situation of an asthma exacerbation (the exacerbation scale; 13 items), the other scale referring to daily life, whenever no exacerbation is present (general scale; 11 items). The CAS has high internal consistency (Cronbach's alpha = .93), excellent test-retest reliability (r = .94), and good construct validity.
Catastrophizing about Asthma Scale | Up to 24 weeks
  In the Catastrophizing about Asthma Scale (CAS) patients rate the extent to which 24 items expressing catastrophic thoughts and feelings about asthma are applicable to themselves (e.g., "There is nothing I can do to reduce the intensity of the asthma attack", "I worry all the time about whether the asthma attack will end", "I feel I can't go on"). The scale has two subscales, one referring to the situation of an asthma exacerbation (the exacerbation scale; 13 items), the other scale referring to daily life, whenever no exacerbation is present (general scale; 11 items). The CAS has high internal consistency (Cronbach's alpha = .93), excellent test-retest reliability (r = .94), and good construct validity.
Latency and summation | Baseline
  In each testing session two series of contacts of the mechanical probe with the flexor digitorum muscle (one at ISI 3 s and one at ISI 5 s) were presented to each forearm. The forearms were always alternated between each series of contacts. Ratings of both forearms were used to control for differences in hand dominance and sites of pain.
Latency and summation | Up to 24 weeks
  In each testing session two series of contacts of the mechanical probe with the flexor digitorum muscle (one at ISI 3 s and one at ISI 5 s) were presented to each forearm. The forearms were always alternated between each series of contacts. Ratings of both forearms were used to control for differences in hand dominance and sites of pain.
Fatigue | Baseline
  Fatigue was measured by the Fatigue Severity Scale. The Fatigue Severity Scale (FSS) was used to assess fatigue and is a 9-item scale, scored from 1 to 7, with the greater the number suggesting more severe fatigue.
Fatigue | Up to 24 weeks
  Fatigue was measured by the Fatigue Severity Scale. The Fatigue Severity Scale (FSS) was used to assess fatigue and is a 9-item scale, scored from 1 to 7, with the greater the number suggesting more severe fatigue.
Health status | Baseline
  The EQ-5D was used to evaluate self-perceived health status and is divided into two sections. The first section contains five questions about mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each question, problems within the domain are evaluated on a three-level basis. Responders can choose between Bno problems^, Bsome problems^, or Bextreme problems^. The second part is a VAS score, which records the responder's self-evaluated health, where 0 is the worst imaginable health and 100 is the best imaginable health.
Health status | Up to 24 weeks
  The EQ-5D was used to evaluate self-perceived health status and is divided into two sections. The first section contains five questions about mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each question, problems within the domain are evaluated on a three-level basis. Responders can choose between Bno problems^, Bsome problems^, or Bextreme problems^. The second part is a VAS score, which records the responder's self-evaluated health, where 0 is the worst imaginable health and 100 is the best imaginable health.
Exercise capacity | Baseline
  The 6MWT is a useful measure of functional capacity, targeted at people with at least moderately severe impairment. It has been widely used for measuring the response to therapeutic interventions for pulmonary and cardiac disease
Exercise capacity | Up to 24 weeks
  The 6MWT is a useful measure of functional capacity, targeted at people with at least moderately severe impairment. It has been widely used for measuring the response to therapeutic interventions for pulmonary and cardiac disease
Kinesiophobia | Baseline
  Kinesiophobia was assessed by the Tampa Scale for Kinesiophobia which evaluate the fear of movement due to dyspnea.
Kinesiophobia | Up to 24 weeks
  Kinesiophobia was assessed by the Tampa Scale for Kinesiophobia which evaluate the fear of movement due to dyspnea.